CLINICAL TRIAL: NCT04232943
Title: A Phase 1 Randomized Study to Examine the Safety, Tolerability, and Immunogenicity of Inactivated Poliovirus Vaccine (IPV) With or Without E.Coli Double Mutant Heat Labile Toxin (dmLT) and Impact on Poliovirus Shedding Post-bOPV Challenge in Healthy IPV-Primed Adult Subjects
Brief Title: Inactivated Poliovirus Vaccine (IPV) With or Without E.Coli Double Mutant Heat-Labile Toxin (dmLT) Challenge Study in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PATH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CVIA 065; 2019-002415-25 (EudraCT Number)
Record Dates: First submitted 2020-01-13; First posted 2020-01-18 (Actual); Results first posted 2022-09-06 (Actual); Last update posted 2022-09-06 (Actual); Status verified 2022-01

CONDITIONS: Polio
Keywords: inactivated polio vaccine (IPV); double mutant [LT(R192G/L211A)] Enterotoxigenic E coli heat toxin (dmLT)
MeSH Terms: conditions — Poliomyelitis | interventions — Poliovirus Vaccine, Inactivated; Adjuvants, Pharmaceutic

STUDY DESIGN:
Intervention Model Description: Participants will receive a single dose of licensed trivalent IPV, administered intramuscularly (IM), with or without dmLT, or bOPV, administered orally (PO). IPV or IPV + dmLT will be administered to groups of 30 participants each. Both participants and clinical staff will be blinded to group assignment (IPV alone vs IPV + dmLT). A positive unblinded control group will be included, composed of 20 participants receiving bOPV. One month (28 days) after receiving study vaccine, all participants will receive a standard oral dose of bOPV to assess relative impact of study vaccine on shedding of that challenge virus.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The study vaccine for Groups 1 and 2 (IPV alone and IPV + dmLT) will be administered IM in a blinded fashion. An unblinded positive control group (Group 3) will be administered bOPV.
  The unblinded Research Pharmacist will perform all preparations of the study product for Groups 1 and 2. Preparation of the study product and administration to the subjects will occur in separate locations to preserve the blinding of staff except for Research Pharmacist. The study subjects, the study personnel who perform study assessments after administration of study product, data entry personnel at the site, and laboratory personnel performing immunologic assays will be blinded to the treatment assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Inactivated Poliomyelitis Vaccine (IPV) (Active Comparator): Participants will receive a single intramuscular injection of 0.5 mL inactivated poliomyelitis vaccine (IPV) on Day 1 followed by a single dose (2 drops) of bivalent oral polio vaccine (bOPV) 28 days later.
  Interventions: Biological: Inactivated Poliomyelitis Vaccine (IPV); Biological: Bivalent Oral Polio Vaccine (bOPV)
- Inactivated Poliomyelitis Vaccine + dmLT (Experimental): Participants will receive a single intramuscular injection of 0.5 mL IPV co-administered with 0.5 μg of dmLT on Day 1 followed by a single dose (2 drops) of bOPV 28 days later.
  Interventions: Biological: Inactivated Poliomyelitis Vaccine (IPV); Biological: E.coli Double Mutant Heat-Labile Toxin (dmLT) (adjuvant); Biological: Bivalent Oral Polio Vaccine (bOPV)
- Bivalent Oral Polio Vaccine (Active Comparator): Participants will receive one dose (2 drops) of bOPV on Day 1 followed by a second dose of bOPV 28 days later.
  Interventions: Biological: Bivalent Oral Polio Vaccine (bOPV)

INTERVENTIONS:
Biological: Inactivated Poliomyelitis Vaccine (IPV) — IMOVAX® Polio is a highly purified, inactivated poliovirus vaccine. Each 0.5 mL dose contains:
  * Type 1 (Mahoney) 40 D-antigen units
  * Type 2 (MEF1) 8 D-antigen units
  * Type 3 (Saukett) 32 D-antigen units
  Other Names: IMOVAX® Polio Vaccine
  Arms: Inactivated Poliomyelitis Vaccine (IPV); Inactivated Poliomyelitis Vaccine + dmLT
Biological: E.coli Double Mutant Heat-Labile Toxin (dmLT) (adjuvant) — LT (R192G/L211A), or "dmLT," is a protein toxoid derived from wild-type enterotoxigenic Escherichia coli (ETEC) labile toxin (LT). The LT toxin has been shown to have inherent mucosal adjuvant properties for co-administered antigens and thus has potential as a mucosal adjuvant for different co-administered vaccines. LT has been genetically modified by replacing the arginine at amino acid position 192 with glycine and the leucine at amino acid position 211 with alanine. These two amino acid substitutions take place in proteolytic cleavage sites, which are critical for activation of the secreted toxin molecules.
  Other Names: LT (R192G/L211A)
  Arms: Inactivated Poliomyelitis Vaccine + dmLT
Biological: Bivalent Oral Polio Vaccine (bOPV) — Polio Sabin™ One and Three (oral) is a bivalent, live attenuated poliomyelitis virus vaccine of the Sabin strains Type 1 (LSc, 2ab) and Type 3 (Leon 12a, 1b), propagated in MRC5 human diploid cells.
  Each dose (0.1 mL) contains not less than 10⁶ 50% cell culture infectious dose (CCID₅₀) of Type 1 and 10⁵·⁸ CCID₅₀ of Type 3.
  Other Names: Polio Sabin™ One and Three (Oral)

SUMMARY:
In this study, the safety and tolerability of inactivated polio vaccine (IPV) co-administered with dmLT will be assessed, as well as whether co-administration of dmLT with IPV enhances mucosal responses compared to those with IPV alone.

DETAILED DESCRIPTION:
A major component of the strategy aimed at worldwide eradication of polio advanced by the World Health Organization (WHO) is based on the replacement of oral polio vaccine (OPV) with IPV; however, IPV is not efficient in preventing person-to-person poliovirus transmission, particularly in settings of poor hygiene, due to limited impact on intestinal mucosal immunity compared to OPV. The addition of an adjuvant, in particular one that may direct the response towards mucosal homing may offset that deficiency.

In this study, the safety and tolerability of IPV co-administered with dmLT will be assessed, as well as whether co-administration of dmLT with IPV enhances mucosal responses to polioviruses types 1, 2, and 3 in comparison with administration of IPV alone and provides greater mucosal immunity, assessed following oral bOPV challenge. The positive control arm (bOPV) is included in order to confirm the level of shedding observable following a dose of an oral vaccine known to develop intestinal immunity.

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female, ages 18-45, inclusive
* Healthy as defined by absence of clinically significant medical condition, either acute or chronic, as determined by medical history and clinical assessment
* History of prior receipt of at least 3 doses of IPV
* Willing and able to provide written informed consent and willing to comply with study requirements
* Intention to remain in the area during the study period
* If female and of childbearing potential, not breastfeeding and not pregnant (based on a negative serum pregnancy test at screening and negative urine pregnancy tests prior to vaccine administration and bOPV challenge), planning to avoid pregnancy until at least three months after bOPV challenge, and willing to use an adequate method of contraception consistently. Effective methods include intrauterine device or hormonal contraceptives (oral, injectable, patch, implant, vaginal ring). Women with credible history of abstinence or in monogamous relationship with a vasectomized partner are also eligible.

Exclusion Criteria:

* History of receiving any OPV at any time
* Receipt of IPV in the last five years
* History of or planned household contact with an individual receiving OPV in prior 4 weeks, or at any point during the study
* Regular contact with children younger than six months (and thus not yet fully vaccinated against polio) and immunocompromised individuals
* Presence of fever on the day of vaccination (oral temperature ≥ 38°C)
* Received an investigational product within 30 days prior to randomization or planning to participate in another research study involving investigational product during the conduct of this study
* Presence of any systemic disorder (cardiovascular, pulmonary, hepatic, renal, gastrointestinal, hematological, endocrine, immunological, dermatological, neurological, cancer or autoimmune diseases) as determined by medical history and/or physical examination that would compromise the participant's health or is likely to result in nonconformance to the protocol or would interfere with the evaluation of responses according to the opinion of the investigator
* History of allergic disease or known hypersensitivity to any component of the study vaccine
* History of anaphylactic reaction
* Receipt of any immunoglobulin therapy and/or blood products in the last 6 months or planned administration during the study period
* History of chronic administration (defined as more than 14 days) of immunosuppressant medications, including oral steroids, parenteral steroids, or high-dose inhaled steroids (> 800 μg/day of beclomethasone dipropionate or equivalent), in the last 6 months to either the study subject or their close household contacts (those on nasal or topical steroids may be permitted to participate in the study)
* Symptoms of an acute self-limited illness, such as an upper respiratory infection or gastroenteritis, including a temperature ≥ 38.0°C, within the 7 days prior to study vaccines administration
* Positive test for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg) or hepatitis C virus (HCV) antibody
* Clinically significant screening laboratory value
* History of receipt of experimental E. coli, enterotoxigenic E. coli (ETEC) labile toxin (LT), or cholera vaccines or live E. coli or Vibrio cholerae challenges.
* Receipt of any licensed vaccine within 28 days before enrollment in this study or plans to receive any licensed vaccine between enrollment and 28 days after the bOPV challenge
* History of alcohol or drug abuse in the last 5 years
* Any condition that in the opinion of the investigator would pose a health risk to the subject if enrolled, or could interfere with the evaluation of the study vaccine

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 87 (Actual)
Dates: Start 2020-01-22 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-02-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Antwerpen, Antwerp, Wilrijk, Belgium

REFERENCES:
- [Derived] Erdem R, De Coster I, Withanage K, Mercer LD, Marchant A, Taton M, Cools N, Lion E, Cassels F, Higgins D, Ivinson K, Locke E, Mahmood K, Wright PF, Gast C, White JA, Ackerman ME, Konopka-Anstadt JL, Mainou BA, Van Damme P. Safety, tolerability, and immunogenicity of inactivated poliovirus vaccine with or without E.coli double mutant heat-labile toxin (dmLT) adjuvant in healthy adults; a phase 1 randomized study. Vaccine. 2023 Mar 3;41(10):1657-1667. doi: 10.1016/j.vaccine.2023.01.048. Epub 2023 Feb 4. PMID 36746739

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at a single center at the University of Antwerp in Belgium.
Pre-assignment Details: Participants were randomized in a 3:3:2 ratio to receive either a single, intramuscular (IM) dose of inactivated poliovirus vaccine (iPV), a single, standard dose of IPV co-administered with a 0.5 μg dose of E.coli double mutant heat-labile toxin (dmLT) or a single oral dose of bivalent oral polio vaccine (bOPV). Twenty-eight (28) days after receiving study vaccine, participants in all groups received a standard oral dose of bOPV challenge.
Groups:
- Inactivated Poliomyelitis Vaccine: Participants received a single intramuscular injection of 0.5 mL inactivated poliomyelitis vaccine (IPV) on Day 1 followed by a single dose (2 drops) of bivalent oral polio vaccine (bOPV) 28 days later.
- Inactivated Poliomyelitis Vaccine + dmLT: Participants received a single intramuscular injection of 0.5 mL IPV co-administered with 0.5 μg of dmLT on Day 1 followed by a single dose (2 drops) of bOPV 28 days later.
- Bivalent Oral Polio Vaccine: Participants received one dose (2 drops) of bOPV on Day 1 followed by a second dose of bOPV 28 days later.
Period: Overall Study
Arm/Group | Inactivated Poliomyelitis Vaccine | Inactivated Poliomyelitis Vaccine + dmLT | Bivalent Oral Polio Vaccine
Started | 32 | 33 | 22
Received Study Vaccination | 30 | 30 | 20
Received bOPV Challenge on Day 29 | 29 | 30 | 20
Completed | 29 | 29 | 20
Not Completed | 3 | 4 | 2
Not completed — Enrolled but Treatment not Administered | 2 | 3 | 2
Not completed — Withdrawal by Subject | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Inactivated Poliomyelitis Vaccine: Participants received a single intramuscular injection of 0.5 mL IPV on Day 1 followed by a single dose (2 drops) of bOPV 28 days later.
- Total: Total of all reporting groups
Arm/Group | Inactivated Poliomyelitis Vaccine | Inactivated Poliomyelitis Vaccine + dmLT | Bivalent Oral Polio Vaccine | Total
Number analyzed (Participants) | 30 | 30 | 20 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 18.9 (1.61) | 18.8 (1.35) | 20.1 (4.18) | 19.2 (2.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 17 | 13 | 48
  Male | 12 | 13 | 7 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 30 | 29 | 19 | 78
  Unknown or Not Reported | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
  Black or African American | 2 | 0 | 1 | 3
  White | 28 | 30 | 18 | 76
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Serious Adverse Events Over the Course of the Study
Description: A serious adverse event (SAE) was any event that resulted in any of the following outcomes:
  1. Death;
  2. Was life-threatening;
  3. Required inpatient hospitalization or prolongation of existing hospitalization;
  4. Resulted in persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions;
  5. Congenital abnormality or birth defect;
  6. Important medical event that did not result in one of the above outcomes but jeopardized the health of the study participant or required medical or surgical intervention to prevent one of the outcomes listed in the above definition of SAE.
Time Frame: Up to 6 months
Population: The total vaccinated population includes all participants in the enrolled population who were randomized and received a study vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | Inactivated Poliomyelitis Vaccine | Inactivated Poliomyelitis Vaccine + dmLT | Bivalent Oral Polio Vaccine
Number analyzed (Participants) | 30 | 30 | 20
Participants | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Severe Adverse Events During the 28 Days Following Study Vaccination
Description: Severe adverse events are events that interrupted a participant's usual daily activity and may have required systemic drug therapy or other treatment. Severe events are usually potentially life-threatening or incapacitating.
Time Frame: Up to 28 days after study vaccination (prior to bOPV challenge)
Population: Total vaccinated population
Measure: Count of Participants; unit: Participants
Arm/Group | Inactivated Poliomyelitis Vaccine | Inactivated Poliomyelitis Vaccine + dmLT | Bivalent Oral Polio Vaccine
Number analyzed (Participants) | 30 | 30 | 20
Participants | 2 | 2 | 0

3. Primary Outcome: Number of Participants With Solicited Local Adverse Events
Description: Solicited adverse events (AEs) are pre-specified local and systemic adverse events that are common or known to be associated with vaccination and that are actively monitored as indicators of vaccine reactogenicity.
  Local/injection site reactions included pain, erythema/redness, swelling, induration, and hyperpigmentation, applicable to participants in the IPV and IPV + dmLT arms who received study injections.
  Severity was graded according to the following:
  Mild: Transient or mild discomfort; does not interfere with activities, erythema or swelling 2.5 - 5 cm, hyperpigmentation 1- 4 cm.
  Moderate: Mild to moderate limitation in activity; no or minimal medical intervention/therapy required, erythema or swelling 5.1 - 10 cm, hyperpigmentation 4.1 - 8 cm, or repeated use of nonnarcotic pain reliever > 24 hours.
  Severe: All normal activity is prevented for 24 hours or more, erythema or swelling > 10 cm, hyperpigmentation > 8 cm, or any use of narcotic pain reliever.
Time Frame: 7 days following study vaccination
Population: Total vaccinated population - participants who received intramuscular injection
Measure: Count of Participants; unit: Participants
Arm/Group | Inactivated Poliomyelitis Vaccine | Inactivated Poliomyelitis Vaccine + dmLT | Bivalent Oral Polio Vaccine
Number analyzed (Participants) | 30 | 30 | 0
Participants
  Mild | 17 | 23 |
  Moderate | 3 | 1 |
  Severe | 0 | 0 |

4. Primary Outcome: Number of Participants With Solicited Systemic Adverse Events
Description: Systemic reactions included fever (oral temperature ≥ 38.0°C), chills, fatigue, headache, muscle aches/myalgia, joint ache/arthralgia, rash, nausea, vomiting, and diarrhea.
  Severity was graded according to the following:
  Mild: Transient or mild discomfort; does not interfere with activities, 2-3 vomiting episodes in 24 hours, 3-5 loose stools/day or diarrhea volume <1000 mL/day, or temperature 38.0 - 38.9˚C.
  Moderate: Mild to moderate limitation in activity; no or minimal medical intervention/therapy required, 4-5 vomiting episodes in 24 hours, 6-9 loose stools/day or 1000-1999 mL output per 24 hours, or temperature 39.0 - 39.9˚C.
  Severe: All normal activity is prevented for 24 hours or more, > 6 vomiting episodes in 24 hours, > 10 loose stools/day or orthostatic hypotension, or temperature > 40.0˚C.
Time Frame: 7 days following study vaccination
Population: Total vaccinated population
Measure: Count of Participants; unit: Participants
Arm/Group | Inactivated Poliomyelitis Vaccine | Inactivated Poliomyelitis Vaccine + dmLT | Bivalent Oral Polio Vaccine
Number analyzed (Participants) | 30 | 30 | 20
Participants
  Mild | 13 | 9 | 9
  Moderate | 4 | 6 | 4
  Severe | 0 | 1 | 0

5. Primary Outcome: Number of Participants With Unsolicited Adverse Events During the 28 Days Following Study Vaccination
Description: An adverse event is any untoward medical occurrence in a participant after administration of the investigational vaccine and that does not necessarily have a causal relationship with the investigational vaccine.
  AEs were graded for severity on the following scale:
  Grade 1 - Mild: Transient or mild discomfort; does not interfere with activities;
  Grade 2 - Moderate: Mild to moderate limitation in activity; no or minimal medical intervention/therapy required;
  Grade 3 - Severe: All normal activity is prevented for 24 hours or more.
Time Frame: 28 days following study vaccination
Population: Total vaccinated population
Measure: Count of Participants; unit: Participants
Arm/Group | Inactivated Poliomyelitis Vaccine | Inactivated Poliomyelitis Vaccine + dmLT | Bivalent Oral Polio Vaccine
Number analyzed (Participants) | 30 | 30 | 20
Participants
  Any adverse event | 14 | 15 | 10
  Severe adverse events | 2 | 2 | 0
  Any adverse event ≥ Grade 2 | 7 | 9 | 4
  Any AE leading to withdrawal | 0 | 0 | 0
  Any adverse event related to study treatment | 5 | 4 | 5

6. Primary Outcome: Percentage of Participants Positive for bOPV Viral Shedding 7 Days Following bOPV Challenge
Description: The presence of the bOPV virus (Sabin strains Type 1 and Type 3) in stool samples was determined using polymerase chain reaction (PCR).
Time Frame: Day 36 (7 days after bOPV challenge)
Population: Participants in the per protocol population who received the bOPV challenge and had available shedding data.
  The per protocol (PP) population includes all enrolled participants who were randomized, received a study vaccination, and who had no protocol violations determined to potentially interfere with the immunogenicity assessment up to each time point.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Inactivated Poliomyelitis Vaccine | Inactivated Poliomyelitis Vaccine + dmLT | Bivalent Oral Polio Vaccine
Number analyzed (Participants) | 28 | 24 | 20
percentage of participants
  Poliovirus Type 1 | 35.7 [18.64 to 55.93] | 41.7 [22.11 to 63.36] | 35.0 [15.39 to 59.22]
  Poliovirus Type 3 | 64.3 [44.07 to 81.36] | 62.5 [40.59 to 81.20] | 40.0 [19.12 to 63.95]
Statistical Analysis 1: Comparison: Inactivated Poliomyelitis Vaccine vs Inactivated Poliomyelitis Vaccine + dmLT; Analysis of Shedding of Poliovirus Type 1; Test type: Other — This study was designed to provide at least 96% power to detect ≥ 60% reduction in shedding rate in the IPV+ dmLT group assuming the shedding rate in the IPV alone group is at least 80%; Risk Ratio (RR) = 1.17, 95% CI 2-sided [0.560 to 2.464] — RR = Ratio of proportions: (IPV+dmLT) / IPV
Statistical Analysis 2: Comparison: Inactivated Poliomyelitis Vaccine vs Inactivated Poliomyelitis Vaccine + dmLT; Analysis of Shedding of Poliovirus Type 3; Test type: Other — [test comment as in outcome 6, analysis 1]; Risk Ratio (RR) = 0.97, 95% CI 2-sided [0.606 to 1.510] — RR = Ratio of proportions: (IPV+dmLT) / IPV

7. Secondary Outcome: Percentage of Participants With a Positive Poliovirus Fecal Neutralization Response 28 Days After Vaccination and 14 Days After bOPV Challenge
Description: Positive response is defined as a minimum 4-fold increase from the pre-vaccination (Baseline) value in fecal anti-poliovirus neutralization antibodies. Serotype-specific poliovirus neutralizing antibody quantitation was conducted using standardized assays at the Wright Laboratory at Dartmouth University.
Time Frame: Day 29 (28 days after study vaccination) and Day 43 (14 days after bOPV challenge)
Population: The per protocol (PP) population includes all enrolled participants who were randomized and received a study vaccination and who had no protocol violations determined to potentially interfere with the immunogenicity assessment up to each time point.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Inactivated Poliomyelitis Vaccine | Inactivated Poliomyelitis Vaccine + dmLT | Bivalent Oral Polio Vaccine
Number analyzed (Participants) | 29 | 26 | 20
percentage of participants
  Serotype 1: Day 29 | 3.4 [0.09 to 17.76] | 0 [0 to 13.23] | 0 [0 to 16.84]
  Serotype 1: Day 43: number analyzed (Participants) | 28 | 24 | 20
  Serotype 1: Day 43 | 3.6 [0.09 to 18.35] | 0 [0 to 14.25] | 0 [0 to 16.84]
  Serotype 2: Day 29 | 0 [0 to 11.94] | 0 [0 to 13.23] | 0 [0 to 16.84]
  Serotype 2: Day 43: number analyzed (Participants) | 28 | 24 | 20
  Serotype 2: Day 43 | 3.6 [0.09 to 18.35] | 0 [0 to 14.25] | 0 [0 to 16.84]
  Serotype 3: Day 29 | 0 [0 to 11.94] | 0 [0 to 13.23] | 0 [0 to 16.84]
  Serotype 3: Day 43: number analyzed (Participants) | 28 | 24 | 20
  Serotype 3: Day 43 | 3.6 [0.09 to 18.35] | 0 [0 to 14.25] | 0 [0 to 16.84]

8. Secondary Outcome: Level of Fecal Poliovirus Immunoglobulin A (IgA) Antibodies at Baseline, 28 Days After Vaccination and 14 Days After bOPV Challenge
Description: Fecal IgA were quantified using a Luminex assay in which monovalent IPVs are covalently conjugated to fluorescently coated beads in order to quantify total and polio-type specific concentrations of IgA in stool specimens.
Time Frame: Baseline (before vaccination), Day 29 (28 days after study vaccination, prior to bOPV challenge) and Day 43 (14 days after bOPV challenge)
Population: Per protocol population with available data at each time point
Measure: Median (95% Confidence Interval); unit: relative fluorescence units
Arm/Group | Inactivated Poliomyelitis Vaccine | Inactivated Poliomyelitis Vaccine + dmLT | Bivalent Oral Polio Vaccine
Number analyzed (Participants) | 30 | 27 | 20
relative fluorescence units
  Serotype 1: Baseline | 4.40 [0.200 to 18.150] | 14.40 [4.900 to 26.900] | 8.65 [1.150 to 16.150]
  Serotype 1: Day 29: number analyzed (Participants) | 29 | 26 | 20
  Serotype 1: Day 29 | 7.60 [1.400 to 13.600] | 1.40 [0.000 to 4.900] | 0.45 [0.000 to 6.400]
  Serotype 1: Day 43: number analyzed (Participants) | 28 | 24 | 20
  Serotype 1: Day 43 | 9.75 [6.100 to 20.100] | 7.60 [1.100 to 17.600] | 3.60 [0.700 to 13.000]
  Serotype 2: Baseline | 13.35 [4.350 to 19.100] | 15.10 [9.100 to 22.100] | 14.10 [6.600 to 32.100]
  Serotype 2: Day 29: number analyzed (Participants) | 29 | 26 | 20
  Serotype 2: Day 29 | 6.10 [3.300 to 17.100] | 8.35 [2.100 to 13.600] | 5.10 [0.050 to 13.600]
  Serotype 2: Day 43: number analyzed (Participants) | 28 | 24 | 20
  Serotype 2: Day 43 | 7.20 [2.650 to 14.300] | 2.80 [0.000 to 11.800] | 3.55 [0.000 to 8.200]
  Serotype 3: Baseline | 13.15 [5.900 to 23.400] | 10.90 [5.900 to 16.400] | 7.90 [0.200 to 20.650]
  Serotype 3: Day 29: number analyzed (Participants) | 29 | 26 | 20
  Serotype 3: Day 29 | 9.40 [1.900 to 15.400] | 3.40 [0.000 to 7.900] | 9.85 [1.900 to 17.900]
  Serotype 3: Day 43: number analyzed (Participants) | 28 | 24 | 20
  Serotype 3: Day 43 | 14.05 [6.800 to 18.300] | 9.10 [2.300 to 13.300] | 8.85 [2.900 to 13.350]

9. Secondary Outcome: Change From Baseline in Fecal Poliovirus IgA Antibodies 28 Days After Study Vaccination and 14 Days After bOPV Challenge
Time Frame: Baseline, Day 29 (28 days after study vaccination, prior to bOPV challenge) and Day 43 (14 days after bOPV challenge)
Population: Per protocol population with available data at each time point
Measure: Median (95% Confidence Interval); unit: relative fluorescence units
Arm/Group | Inactivated Poliomyelitis Vaccine | Inactivated Poliomyelitis Vaccine + dmLT | Bivalent Oral Polio Vaccine
Number analyzed (Participants) | 29 | 26 | 20
relative fluorescence units
  Serotype 1: Day 29 | 0.00 [-5.000 to 7.600] | -7.90 [-21.200 to -3.700] | -2.95 [-10.200 to 1.450]
  Serotype 1: Day 43: number analyzed (Participants) | 28 | 24 | 20
  Serotype 1: Day 43 | 3.05 [0.000 to 9.500] | -8.60 [-14.400 to 0.200] | -1.65 [-9.900 to 0.100]
  Serotype 2: Day 29 | 0.00 [-8.300 to 3.500] | -3.75 [-14.650 to 1.850] | -11.75 [-23.050 to -0.550]
  Serotype 2: Day 43: number analyzed (Participants) | 28 | 24 | 20
  Serotype 2: Day 43 | 0.00 [-9.550 to 1.000] | -9.35 [-15.300 to 0.000] | -14.10 [-28.100 to -2.950]
  Serotype 3: Day 29 | -0.50 [-10.400 to 4.900] | -4.00 [-11.000 to -0.950] | -0.20 [-11.500 to 5.900]
  Serotype 3: Day 43: number analyzed (Participants) | 28 | 24 | 20
  Serotype 3: Day 43 | 4.80 [-4.100 to 12.400] | -3.25 [-6.900 to 5.400] | -0.20 [-15.600 to 8.100]

10. Secondary Outcome: Serum Neutralizing Antibody Seroconversion Rate 28 Days After Study Vaccination
Description: Serum neutralizing antibody seroconversion rate is defined as the percentage of participants demonstrating a minimum four-fold increase in type-specific poliovirus serum neutralizing antibody titers between baseline and 28 days post vaccination, or post-vaccination titer > 1:8 if seronegative at baseline.
Time Frame: Day 29 (28 days after study vaccination, prior to bOPV challenge)
Population: Per protocol population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Inactivated Poliomyelitis Vaccine | Inactivated Poliomyelitis Vaccine + dmLT | Bivalent Oral Polio Vaccine
Number analyzed (Participants) | 29 | 25 | 20
percentage of participants
  Serotype 1 | 93.1 [77.23 to 99.15] | 84.0 [63.92 to 95.46] | 80.0 [56.34 to 94.27]
  Serotype 2 | 100 [88.06 to 100] | 92.0 [73.97 to 99.02] | 15.0 [3.21 to 37.89]
  Serotype 3 | 86.2 [68.34 to 96.11] | 96.0 [79.65 to 99.90] | 50.0 [27.20 to 72.80]

11. Secondary Outcome: Geometric Mean Titer of Serum Poliovirus Neutralizing Antibodies at Baseline and 28 Days After Study Vaccination
Time Frame: Baseline (pre-vaccination) and Day 29 (28 days after study vaccination, prior to bOPV challenge)
Population: Per protocol population with available data at each time point
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Inactivated Poliomyelitis Vaccine | Inactivated Poliomyelitis Vaccine + dmLT | Bivalent Oral Polio Vaccine
Number analyzed (Participants) | 30 | 27 | 20
titer
  Serotype 1: Baseline | 190.5 [110.19 to 329.43] | 422.7 [238.89 to 747.83] | 248.7 [128.91 to 479.70]
  Serotype 1: Day 29: number analyzed (Participants) | 29 | 25 | 20
  Serotype 1: Day 29 | 18731 [10502 to 33405] | 25048 [13152 to 47705] | 15657 [7770.3 to 31549]
  Serotype 2: Baseline | 187.9 [93.36 to 378.07] | 205.0 [100.47 to 418.37] | 221.2 [96.30 to 508.11]
  Serotype 2: Day 29: number analyzed (Participants) | 29 | 25 | 20
  Serotype 2: Day 29 | 45241 [24760 to 82665] | 43251 [23053 to 81147] | 241.3 [119.95 to 485.51]
  Serotype 3: Baseline | 1021.6 [554.63 to 1881.9] | 1266.4 [666.45 to 2406.4] | 2041.3 [956.82 to 4354.9]
  Serotype 3: Day 29: number analyzed (Participants) | 29 | 25 | 20
  Serotype 3: Day 29 | 91419 [55229 to 151324] | 52165 [30175 to 90179] | 7874.5 [4331.6 to 14315]

12. Secondary Outcome: Seroprotection Rate of Serum Poliovirus Neutralizing Antibodies at Baseline and 28 Days Following Vaccination
Description: Seroprotection rate of serum poliovirus neutralizing antibodies is defined as a type-specific poliovirus serum neutralizing antibody titer ≥ 1:8.
Time Frame: Baseline (before vaccination) and Day 29 (28 days after vaccination, prior to bOPV challenge)
Population: Per protocol population with available data at each time point
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Inactivated Poliomyelitis Vaccine | Inactivated Poliomyelitis Vaccine + dmLT | Bivalent Oral Polio Vaccine
Number analyzed (Participants) | 30 | 27 | 20
percentage of participants
  Serotype 1: Baseline | 93.3 [77.93 to 99.18] | 100 [87.23 to 100] | 100 [83.16 to 100]
  Serotype1: Day 29: number analyzed (Participants) | 29 | 25 | 20
  Serotype1: Day 29 | 100 [88.06 to 100] | 100 [86.28 to 100] | 100 [83.16 to 100]
  Serotype 2: Baseline | 93.3 [77.93 to 99.18] | 96.3 [81.03 to 99.91] | 90.0 [68.30 to 98.77]
  Serotype 2: Day 29: number analyzed (Participants) | 29 | 25 | 20
  Serotype 2: Day 29 | 100 [88.06 to 100] | 100 [86.28 to 100] | 95.0 [75.13 to 99.87]
  Serotype 3: Baseline | 100 [88.43 to 100] | 100 [87.23 to 100] | 90.0 [68.30 to 98.77]
  Serotype 3: Day 29: number analyzed (Participants) | 29 | 25 | 20
  Serotype 3: Day 29 | 100 [88.06 to 100] | 100 [86.28 to 100] | 100 [83.16 to 100]

13. Secondary Outcome: Geometric Mean Fold-Rise in Serum Poliovirus Neutralizing Antibodies
Time Frame: Baseline (before vaccination) and Day 29 (28 days after vaccination, prior to bOPV challenge)
Population: Per protocol population
Measure: Geometric Mean (95% Confidence Interval); unit: fold-rise
Arm/Group | Inactivated Poliomyelitis Vaccine | Inactivated Poliomyelitis Vaccine + dmLT | Bivalent Oral Polio Vaccine
Number analyzed (Participants) | 29 | 25 | 20
fold-rise
  Serotype 1 | 134.3 [53.94 to 334.23] | 54.2 [20.27 to 144.98] | 40.8 [13.60 to 122.27]
  Serotype 2 | 346.7 [121.99 to 985.30] | 151.9 [49.54 to 465.86] | 0.8 [0.22 to 2.66]
  Serotype 3 | 103.9 [40.67 to 265.47] | 41.5 [15.09 to 113.85] | 8.6 [2.77 to 26.47]

14. Secondary Outcome: Percentage of Participants With a Circulating Poliovirus IgA Antibody-Secreting Cell Response
Description: Poliovirus antibody secreting cell (ASC) response is defined as ≥ 8 ASC/10⁶ peripheral blood mononuclear cells (PBMC) at any time point following both study vaccination and bOPV challenge.
Time Frame: Baseline (pre-vaccination), Day 8 (7 days after study vaccination), Day 29 (28 days after study vaccination prior to bOPV challenge), and Day 36 (7 days after bOPV challenge)
Population: Per protocol population with available data at each time point
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Inactivated Poliomyelitis Vaccine | Inactivated Poliomyelitis Vaccine + dmLT | Bivalent Oral Polio Vaccine
Number analyzed (Participants) | 30 | 27 | 20
percentage of participants
  Serotype 1: Baseline | 0.0 [0.00 to 11.57] | 0.0 [0.00 to 12.77] | 0.0 [0.00 to 16.84]
  Serotype 1: Day 8 | 10.0 [2.11 to 26.53] | 7.4 [0.91 to 24.29] | 25.0 [8.66 to 49.10]
  Serotype 1: Day 29: number analyzed (Participants) | 29 | 26 | 20
  Serotype 1: Day 29 | 0.0 [0.00 to 11.94] | 0.0 [0.00 to 13.23] | 0.0 [0.00 to 16.84]
  Serotype 1: Day 36: number analyzed (Participants) | 29 | 26 | 20
  Serotype 1: Day 36 | 6.9 [0.85 to 22.77] | 15.4 [4.36 to 34.87] | 0.0 [0.00 to 16.84]
  Serotype 2: Baseline | 0.0 [0.00 to 11.57] | 0.0 [0.00 to 12.77] | 0.0 [0.00 to 16.84]
  Serotype 2: Day 8 | 6.7 [0.82 to 22.07] | 3.7 [0.09 to 18.97] | 10.0 [1.23 to 31.70]
  Serotype 2: Day 29: number analyzed (Participants) | 29 | 26 | 20
  Serotype 2: Day 29 | 0.0 [0.00 to 11.94] | 0.0 [0.00 to 13.23] | 0.0 [0.00 to 16.84]
  Serotype 2: Day 36: number analyzed (Participants) | 29 | 26 | 20
  Serotype 2: Day 36 | 3.4 [0.09 to 17.76] | 7.7 [0.95 to 25.13] | 0.0 [0.00 to 16.84]
  Serotype 3: Baseline | 0.0 [0.00 to 11.57] | 0.0 [0.00 to 12.77] | 0.0 [0.00 to 16.84]
  Serotype 3: Day 8 | 3.3 [0.08 to 17.22] | 3.7 [0.09 to 18.97] | 15.0 [3.21 to 37.89]
  Serotype 3: Day 29: number analyzed (Participants) | 29 | 26 | 20
  Serotype 3: Day 29 | 0.0 [0.00 to 11.94] | 0.0 [0.00 to 13.23] | 0.0 [0.00 to 16.84]
  Serotype 3: Day 36: number analyzed (Participants) | 29 | 26 | 20
  Serotype 3: Day 36 | 3.4 [0.09 to 17.76] | 7.7 [0.95 to 25.13] | 0.0 [0.00 to 16.84]

15. Secondary Outcome: Number of Circulating Poliovirus IgA Antibody Secreting Cells at Baseline and After Study Vaccination
Time Frame: as for outcome 14
Population: Per protocol population with available data at each time point
Measure: Median (95% Confidence Interval); unit: cells/10⁶ PBMC
Arm/Group | Inactivated Poliomyelitis Vaccine | Inactivated Poliomyelitis Vaccine + dmLT | Bivalent Oral Polio Vaccine
Number analyzed (Participants) | 30 | 27 | 20
cells/10⁶ PBMC
  Serotype 1: Baseline | 0.00 [0.000 to 0.250] | 0.00 [0.000 to 0.167] | 0.00 [0.000 to 0.000]
  Serotype 1: Day 8 | 0.17 [0.000 to 0.292] | 0.50 [0.000 to 1.250] | 0.63 [0.000 to 4.917]
  Serotype 1: Day 29: number analyzed (Participants) | 29 | 26 | 20
  Serotype 1: Day 29 | 0.00 [0.000 to 0.000] | 0.00 [0.000 to 0.000] | 0.00 [0.000 to 0.250]
  Serotype 1: Day 36: number analyzed (Participants) | 29 | 26 | 20
  Serotype 1: Day 36 | 0.92 [0.250 to 2.750] | 0.38 [0.000 to 2.500] | 0.17 [0.000 to 0.708]
  Serotype 2: Baseline | 0.00 [0.000 to 0.125] | 0.00 [0.000 to 0.083] | 0.00 [0.000 to 0.333]
  Serotype 2: Day 8 | 0.17 [0.000 to 0.313] | 0.00 [0.000 to 0.750] | 0.00 [0.000 to 0.167]
  Serotype 2: Day 29: number analyzed (Participants) | 29 | 26 | 20
  Serotype 2: Day 29 | 0.00 [0.000 to 0.000] | 0.00 [0.000 to 0.250] | 0.00 [0.000 to 0.250]
  Serotype 2: Day 36: number analyzed (Participants) | 29 | 26 | 20
  Serotype 2: Day 36 | 0.33 [0.000 to 1.250] | 0.08 [0.000 to 0.250] | 0.00 [0.000 to 0.500]
  Serotype 3: Baseline | 0.00 [0.000 to 0.333] | 0.00 [0.000 to 0.000] | 0.21 [0.000 to 0.250]
  Serotype 3: Day 8 | 0.00 [0.000 to 0.083] | 0.00 [0.000 to 0.250] | 0.00 [0.000 to 0.375]
  Serotype 3: Day 29: number analyzed (Participants) | 29 | 26 | 20
  Serotype 3: Day 29 | 0.00 [0.000 to 0.000] | 0.00 [0.000 to 0.000] | 0.00 [0.000 to 0.125]
  Serotype 3: Day 36: number analyzed (Participants) | 29 | 26 | 20
  Serotype 3: Day 36 | 0.25 [0.000 to 0.667] | 0.00 [0.000 to 0.500] | 0.00 [0.000 to 0.375]

16. Secondary Outcome: Percentage of Participants With a Circulating Poliovirus Immunoglobulin G (IgG) Antibody-Secreting Cell Response
Description: as for outcome 14
Time Frame: as for outcome 14
Population: Per protocol population with available data at each time point
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Inactivated Poliomyelitis Vaccine | Inactivated Poliomyelitis Vaccine + dmLT | Bivalent Oral Polio Vaccine
Number analyzed (Participants) | 30 | 27 | 20
percentage of participants
  Serotype 1: Baseline | 0.0 [0.00 to 11.57] | 0.0 [0.00 to 12.77] | 0.0 [0.00 to 16.84]
  Serotype 1: Day 8 | 90.0 [73.47 to 97.89] | 74.1 [53.72 to 88.89] | 50.0 [27.20 to 72.80]
  Serotype 1: Day 29: number analyzed (Participants) | 29 | 26 | 20
  Serotype 1: Day 29 | 0.0 [0.00 to 11.94] | 0.0 [0.00 to 13.23] | 0.0 [0.00 to 16.84]
  Serotype 1: Day 36: number analyzed (Participants) | 29 | 26 | 20
  Serotype 1: Day 36 | 27.6 [12.73 to 47.24] | 23.1 [8.97 to 43.65] | 10.0 [1.23 to 31.70]
  Serotype 2: Baseline | 0.0 [0.00 to 11.57] | 0.0 [0.00 to 12.77] | 0.0 [0.00 to 16.84]
  Serotype 2: Day 8 | 56.7 [37.43 to 74.54] | 51.9 [31.95 to 71.33] | 10.0 [1.23 to 31.70]
  Serotype 2: Day 29: number analyzed (Participants) | 29 | 26 | 20
  Serotype 2: Day 29 | 0.0 [0.00 to 11.94] | 0.0 [0.00 to 13.23] | 0.0 [0.00 to 16.84]
  Serotype 2: Day 36: number analyzed (Participants) | 29 | 26 | 20
  Serotype 2: Day 36 | 3.4 [0.09 to 17.76] | 3.8 [0.10 to 19.64] | 0.0 [0.00 to 16.84]
  Serotype 3: Baseline | 0.0 [0.00 to 11.57] | 0.0 [0.00 to 12.77] | 0.0 [0.00 to 16.84]
  Serotype 3: Day 8 | 40.0 [22.66 to 59.40] | 40.7 [22.39 to 61.20] | 20.0 [5.73 to 43.66]
  Serotype 3: Day 29: number analyzed (Participants) | 29 | 26 | 20
  Serotype 3: Day 29 | 0.0 [0.00 to 11.94] | 0.0 [0.00 to 13.23] | 0.0 [0.00 to 16.84]
  Serotype 3: Day 36: number analyzed (Participants) | 29 | 26 | 20
  Serotype 3: Day 36 | 13.8 [3.89 to 31.66] | 3.8 [0.10 to 19.64] | 5.0 [0.13 to 24.87]

17. Secondary Outcome: Number of Circulating Poliovirus IgG Antibody Secreting Cells at Baseline and After Study Vaccination
Time Frame: as for outcome 14
Population: Per protocol population with available data at each time point
Measure: Median (95% Confidence Interval); unit: cells/10⁶ PBMC
Arm/Group | Inactivated Poliomyelitis Vaccine | Inactivated Poliomyelitis Vaccine + dmLT | Bivalent Oral Polio Vaccine
Number analyzed (Participants) | 30 | 27 | 20
cells/10⁶ PBMC
  Serotype 1: Baseline | 0.25 [0.000 to 0.375] | 0.00 [0.000 to 0.000] | 0.13 [0.000 to 0.500]
  Serotype 1: Day 8 | 29.75 [23.000 to 45.750] | 18.00 [9.750 to 49.500] | 7.00 [1.000 to 19.375]
  Serotype 1: Day 29: number analyzed (Participants) | 29 | 26 | 20
  Serotype 1: Day 29 | 0.00 [0.000 to 0.000] | 0.00 [0.000 to 0.250] | 0.00 [0.000 to 0.000]
  Serotype 1: Day 36: number analyzed (Participants) | 29 | 26 | 20
  Serotype 1: Day 36 | 3.00 [0.750 to 5.000] | 2.00 [0.000 to 5.125] | 0.38 [0.000 to 1.000]
  Serotype 2: Baseline | 0.13 [00000 to 0.375] | 0.25 [0.000 to 0.250] | 0.00 [0.000 to 0.000]
  Serotype 2: Day 8 | 11.13 [5.875 to 20.500] | 9.50 [2.250 to 19.000] | 0.13 [0.000 to 0.250]
  Serotype 2: Day 29: number analyzed (Participants) | 29 | 26 | 20
  Serotype 2: Day 29 | 0.00 [0.000 to 0.000] | 0.00 [0.000 to 0.375] | 0.00 [0.000 to 0.250]
  Serotype 2: Day 36: number analyzed (Participants) | 29 | 26 | 20
  Serotype 2: Day 36 | 0.50 [0.000 to 1.000] | 0.25 [0.000 to 1.375] | 0.00 [0.000 to 0.375]
  Serotype 3: Baseline | 0.00 [0.000 to 0.125] | 0.00 [0.000 to 0.250] | 0.00 [0.000 to 0.250]
  Serotype 3: Day 8 | 5.00 [2.500 to 11.500] | 5.25 [1.500 to 14.750] | 0.25 [0.000 to 4.875]
  Serotype 3: Day 29: number analyzed (Participants) | 29 | 26 | 20
  Serotype 3: Day 29 | 0.00 [0.000 to 0.000] | 0.00 [0.000 to 0.250] | 0.00 [0.000 to 0.000]
  Serotype 3: Day 36: number analyzed (Participants) | 29 | 26 | 20
  Serotype 3: Day 36 | 0.00 [0.000 to 1.000] | 0.50 [0.000 to 1.750] | 0.00 [0.000 to 0.250]

18. Secondary Outcome: Area Under the Curve (AUC) of Viral Shedding in Stool for 28 Days After bOPV Challenge
Description: AUC was calculated using the linear trapezoidal rule with all samples collected from Day 33 to 57.
Time Frame: Days 33, 36, 43, 50, and 57 (i.e., 4, 7, 14, 21, and 28 days, respectively, following bOPV challenge).
Population: Per protocol population
Measure: Median (Standard Deviation); unit: log₁₀(CCID₅₀/g) * days
Arm/Group | Inactivated Poliomyelitis Vaccine | Inactivated Poliomyelitis Vaccine + dmLT | Bivalent Oral Polio Vaccine
Number analyzed (Participants) | 29 | 26 | 20
log₁₀(CCID₅₀/g) * days | 43.578 (25.381) | 46.867 (33.673) | 13.138 (27.627)

19. Secondary Outcome: Time to Cessation of Viral Shedding in Stool After bOPV Challenge
Description: Time to cessation of viral shedding in stool is defined as the study day of the first instance of 3 consecutive samples PCR-negative for virus, with samples taken on separate days.
Time Frame: Days 33, 36, 39, 43, 46, 50, and 57
Population: Per-protocol population participants who received the bOPV challenge and had post-challenge viral shedding results.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Inactivated Poliomyelitis Vaccine | Inactivated Poliomyelitis Vaccine + dmLT | Bivalent Oral Polio Vaccine
Number analyzed (Participants) | 29 | 27 | 20
days
  Poliovirus Type I | 6 [5 to 9] | 7 [5 to 14] | 5 [4 to 9]
  Poliovirus Type 3 | NA [NA to NA] — Could not be estimated due to the low number of events | 19 [10 to 27] | 5 [4 to 11]

ADVERSE EVENTS:
Time Frame: Serious adverse events were collected from first dose up to Day 169 (6 months). Non-serious adverse events were collected up to 28 days after each vaccination.
Arm/Group | Inactivated Poliomyelitis Vaccine | Inactivated Poliomyelitis Vaccine + dmLT | Bivalent Oral Polio Vaccine
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/20
Other Adverse Events (participants affected / at risk) | 29/30 | 28/30 | 15/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Inactivated Poliomyelitis Vaccine (N=30) | Inactivated Poliomyelitis Vaccine + dmLT (N=30) | Bivalent Oral Polio Vaccine (N=20)
Injection site pain (General disorders) | 22 (24) | 24 (24) | 0 (0)
Fatigue (General disorders) | 11 (11) | 13 (16) | 9 (9)
Chills (General disorders) | 0 (0) | 1 (1) | 1 (1)
Injection site induration (General disorders) | 1 (1) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 2 (2) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 1 (1) | 0 (0)
Injection site discolouration (General disorders) | 0 (0) | 1 (1) | 0 (0)
Injection site erythema (General disorders) | 0 (0) | 1 (1) | 0 (0)
Injection site haemorrhage (General disorders) | 0 (0) | 1 (1) | 0 (0)
Injection site swelling (General disorders) | 1 (1) | 0 (0) | 0 (0)
Injection site warmth (General disorders) | 1 (1) | 0 (0) | 0 (0)
Thirst (General disorders) | 1 (1) | 0 (0) | 0 (0)
Vessel puncture site erythema (General disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 15 (16) | 17 (26) | 14 (14)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 4 (5) | 7 (10)
Nausea (Gastrointestinal disorders) | 7 (7) | 5 (6) | 4 (4)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (2) | 3 (3)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Aphthous ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 9 (10) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (2) | 2 (2) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gingivitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pulpitis dental (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 2 (2) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
C-reactive protein increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Excessive cerumen production (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Motion sickness (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Blepharitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Eye irritation (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Allergy to arthropod bite (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-06-03): https://cdn.clinicaltrials.gov/large-docs/43/NCT04232943/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-18): https://cdn.clinicaltrials.gov/large-docs/43/NCT04232943/SAP_001.pdf